CLINICAL TRIAL: NCT02437175
Title: Efficacy of Food Supplements Containing Trace Elements in the Treatment of Endometriosis, Combined or Not to an Adenomyosis: a Pilot Study
Brief Title: Efficacy of Trace Elements in the Treatment of Endometriosis: a Pilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Pronutri (Industry)
Collaborators: Expert Clinical Services Organization (ECSOR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pronutri-IIIa-001
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Endometriosis
Keywords: pelvic pain; quality of life; adenomyosis
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Adenomyosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo: 1 sequence of 10 tablets on the morning and 1 sequence of 10 tablets at the evening, daily, during 120 days.
  Interventions: Dietary Supplement: Placebo
- Trace elements (Experimental): NUTRI ENDO 1 (1 sequence of 10 tablets on the morning) and NUTRI ENDO 2 ( sequence of 10 tablets at the evening), daily, during 120 days.
  Interventions: Dietary Supplement: ENDO 1/ENDO 2

INTERVENTIONS:
Dietary Supplement: ENDO 1/ENDO 2 — NUTRI ENDO 1 (1 sequence of 10 tablets on the morning) and NUTRI ENDO 2 ( sequence of 10 tablets at the evening), daily, during 120 days.
  Arms: Trace elements
Dietary Supplement: Placebo — Placebo: 1 sequence of 10 tablets on the morning and 1 sequence of 10 tablets at the evening, daily, during 120 days.
  Arms: Placebo

SUMMARY:
The primary objective of this pilot study is to evaluate the efficacy of trace elements, versus placebo, on the reduction of pain in endometriosis of an American Fertility Society (AFSr) score of 2 to 4, combined or not to an adenomyosis, during a chronic treatment of 4 months.

DETAILED DESCRIPTION:
The objectives of this pilot study are to evaluate the efficacy of trace elements, versus placebo, on the reduction of pain, on the quality of life, on the use of rescue medication (ibuprofen) in patients with an endometriosis of an American Fertility Society (AFSr) score of 2 to 4, combined or not to an adenomyosis, during a chronic treatment of 4 months. The safety of trace elements versus placebo will also be assessed.

This will be a prospective, interventional, randomized, placebo-controlled, two parallel-group, double-blind study.

Trace elements or placebo are administered in the absence of any other treatment or as add-on treatments to common therapies such as sexual hormones, anti-inflammatory drugs or surgery.

A run-in placebo period of 30 days will allow eliminating the patients who are responding to strongly to a placebo.

The treatment will last for 4 months. The total duration of the study will be 5 months for each patient. Four medical visits (Days -45 to -30, 0, 60 and 120) and two phone contacts (Days 30 and 90) will be scheduled.

A urine pregnancy test will be undertaken at each visit. The quality of life scale (EHP-30) will be filled in on Days 0, 60 and 120. During the whole study period, patients will be asked to fill in a diary, in which they will score their pain on a visual analog scale, their blood loss and their consumption of rescue medication (ibuprofen).

Phone contacts will be used to reinforce the compliance and to collect potential adverse events.

Non-serious and serious adverse events will be collected between Days 0 and 120.

All concomitant medications will be recorded, including the rescue medication between Day -45 and Day 120.

A paper case report form will be used.

A total of 60 patients (30 receiving trace elements and 30 receiving placebo) will be randomized to achieve a total of 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Woman suffering from an AFSr 2 to 4 endometriosis (combined or not to an adenomyosis), confirmed by laparoscopy, laparotomy or MRI as well as by a biopsy (done within 3 years before inclusion in the study), treated or not with sexual hormones, contraceptive or not (stable treatment for minimum 2 months) or any other treatment
* Time period of at least 6 months after surgical treatment
* Age between 18 and 45 years
* Non-menopausal woman
* Baseline pain (Day -45 to -30) of at least 40 mm on a visual analog scale
* No reduction of more than 20% of pain on the visual analog scale after the run-in placebo period.

Exclusion Criteria:

* AFSr 1 endometriosis
* Adenomyosis without endometriosis
* Pregnancy
* Existence of another pathology that could interfere with endometriosis and/or with adenomyosis, and the study follow-up
* Psychological or psychiatric conditions
* Patient who, according to the investigator, will not be able to comply to the prerequisites of the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Pain (visual analog scale) | Day 0 to Day 120
  Pain scored daily by the patient using a visual analog scale

SECONDARY OUTCOMES:
EHP-30 (validated 30-items questionnaire) | Day 0 to Day 120
  Quality of life determined using a validated 30-items questionnaire (EHP-30)
Rescue medication consumption (Number of ibuprofen tablets consumed) | Day 0 to Day 120
Safety (Non-serious and serious adverse events (related or not) | Day 0 to Day 120
  Non-serious and serious adverse events (related or not)

CONTACTS AND LOCATIONS:
Overall Officials: Didier Oberweis, MD, Principal Investigator — CHU Vésale
Locations (1):
- CHU Vésale, Montigny-le-Tilleul, Hainaut, Belgium

REFERENCES:
- See also: A pilot double-blind, randomized, placebo-controlled trial of the efficacy of trace elements in the treatment of endometriosis-related pain: study design and methodology — https://www.dovepress.com/articles.php?article_id=25534
- Available data/document: Methodology paper — https://www.dovepress.com/articles.php?article_id=25534